CLINICAL TRIAL: NCT07152626
Title: Combination Approach With Ritlecitinib and nbUVB Compared to Ritlecitinib Alone for Treating Vitiligo Prospective Multicentric Evaluator Blinded Interventional Study
Brief Title: Combination Approach With Ritlecitinib and nbUVB Compared to Ritlecitinib Alone for Treating Vitiligo
Acronym: COMBIVIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-PP-03; 2025-521504-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug alone (Active Comparator): Patients will be assigned to receive either ritlecitinib 100mg daily (QD)
  Interventions: Drug: LITFULO
- Drug and UVB (Experimental): patients will be assigned to receive a combined therapy using ritlecitinib 100mg QD + twice weekly narrowband UVB treatment for a duration of 52 weeks.
  Interventions: Procedure: LITFULO and UVB

INTERVENTIONS:
Drug: LITFULO — Following central randomization, patients will be assigned to receive either ritlecitinib 100mg daily (QD) or a combined therapy using ritlecitinib 100mg QD + twice weekly narrowband UVB treatment for a duration of 52 weeks. At the end of this period, all participants will continue for the open-label phase, receiving ritlecitinib 100mg QD. Eligible participants will be stratified by Fitzpatrick Skin Type (FST, also known as phototype).
  Arms: Drug alone
Procedure: LITFULO and UVB — Following central randomization, patients will be assigned to receive either ritlecitinib 100mg daily (QD) or a combined therapy using ritlecitinib 100mg QD + twice weekly narrowband UVB treatment for a duration of 52 weeks. At the end of this period, all participants will continue for the open-label phase, receiving ritlecitinib 100mg QD. Eligible participants will be stratified by Fitzpatrick Skin Type (FST, also known as phototype).
  Arms: Drug and UVB

SUMMARY:
Vitiligo affects approximately 1 to 2% of the global population and significantly impacts people's quality of life. areas of high stress. Ritlecitinib, an orally administered inhibitor of JAK3 (Janus kinase)/ TEC (tyrosine kinase expressed in hepatocellular carcinoma) has shown effectiveness and safety for the treatment of vitiligo. In a phase 2b trial, three doses of ritlecitinib, 200/50 mg, 100/50 mg, and 50 mg, were all statistically significant versus placebo on the Facial Vitiligo Area Scoring Index (F-VASI) at week 24 in patients with active NSV. Considering that the immune process primarily contributes to depigmentation while ultraviolet (UV) radiation stimulates the differentiation and proliferation of melanocyte stem cells for re-pigmentation, the investigators propose that a combination therapy using ritlecitinib and narrowband UVB (nbUVB) could offer an optimal approach for treating vitiligo patients.

The primary objective is thTo compare between the groups, the mean percentage change from baseline in F-VASI and T-VASI at week 52.

Following central randomization, patients will be assigned to receive either ritlecitinib 100mg daily (QD) or a combined therapy using ritlecitinib 100mg QD + twice weekly narrowband UVB treatment for a duration of 52 weeks. At the end of this period, all participants will continue for the open-label phase, receiving ritlecitinib 100mg QD. Eligible participants will be stratified by Fitzpatrick Skin Type (FST, also known as phototype). More specifically, there will be 2 strata based on FST targets: (1) FST I to III (2) FST I IV, to VI. Each FST stratum will target to enroll at least 50% participants into the study population. Stratified randomization across FST sub-groups will support the evaluation of a consistent benefit-risk profile across all FST strata. Enrollment of participants with active or stable nonsegmental vitiligo will be proactively managed without formally capping or stratifying.

Throughout the study, there will be a total of 8 visits conducted: selection, inclusion, week 4, week 12, week 24, week 36, week 52 and week 72. In patients who volunteer, a skin biopsy will be performed on both the lesional and perilesional areas at baseline, week 4 and week 52. We aim to include between 12 and 20 volunteer patients. Serum and plasma samples will be collected at the screening visit, week 4, week 12, week 24, week 36, week 52 and week 72.

A pregnancy test will be performed every 4 weeks i.e. at weeks 8, 16, 20, 28, 32, 40, 44, 48, 56, 60, 64 and 68;

ELIGIBILITY:
Inclusion Criteria:

* 1. Men and women with non-segmental vitiligo. 2. Age ≥ 18 age old 3. BSA involvement between 4% and 60% inclusive, excluding involvements at palms of the hands, soles of the feet, or dorsal aspect of the feet 4. BSA ≥0.5% involvement on the face (face is defined as including the area on the forehead to the original hairline, on the cheek vertically to the jawline, and laterally from the corner of the mouth to the tragus. The face will not include scalp, ears, neck, or surface area of the lips, but will include the nose and the eyelids) 5. F-VASI ≥0.5 and T-VASI ≥3 6. Active and stable vitiligo 7. For Women of childbearing potential (WOCBP), an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study; Women of childbearing potential (WOCBP) must have a negative urine pregnancy test result at baseline; WOCBP are defined as women who are biologically capable of becoming pregnant, including women who are using contraceptives or whose sexual partners are either sterile or using contraceptives;

Women of non-childbearing potential (WONCBP) do not require a urine pregnancy test and must meet at least one of the following criteria:

o Have undergone hysterectomy or bilateral oophorectomy;

* Have medically confirmed ovarian failure; or
* Are medically confirmed to be post-menopausal (cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause); 8. Affiliation to a social security system; 9. Signed informed consent.

Exclusion Criteria:

* 1. Pregnant or breast-feeding women. Or women with potential childbearing and not taking contraceptives or who plan to get pregnant during the study duration, and 2. Segmental or mixed vitiligo, and 3. Contraindication to nbUVB phototherapy, and 4. Concomitant use of topical or systemic immunosuppressive medication or steroids, and 5. Patients treated before with oral JAK inhibitor, topical treatments (including JAK inhibitors) that could affect vitiligo (eg, corticosteroids, vitamin D3 and calcineurin inhibitor) within 2 Weeks of Day 1 (Baseline) and during the study

At any time prior to or during the study:

* Use of permanent depigmentation treatment for vitiligo and/or other types of pigmentation disorder (eg, monobenzone or phenol).
* Previous use of any systemic JAK inhibitor for any disease indication
* Any non-B cell selective lymphocyte depleting agent (eg, alefacept, alemtuzumab) and alkylating agents [eg, cyclophosphamide or chlorambucil], total lymphoid irradiation, etc.
* History of MKTP or other surgical treatment for vitiligo.

Within 6 months of the first dose of study drug or 5 half-lives (if known), or until lymphocyte count returns to normal, whichever is longer and during the study:

- Any B-cell-depleting agents including but not limited to rituximab or previously receiving leukocyte apheresis, including selective lymphocyte, monocyte, or granulocyte apheresis, or plasma exchange.

Within 12 weeks of first dose of study drug or 5 half-lives (if known), whichever is longer and during the study:

* Other immunomodulatory biologic agents or other marketed immunosuppressants.
* IL12/23 inhibitor (eg, ustekinumab)
* Integrin inhibitors (eg, vedolizumab)

Within 8 weeks of Day 1 and during the study:

- Narrow-band UVB phototherapy, Psoralen Ultra-Violet A therapy, or other phototherapy.

TNF inhibitors (or biosimilars thereof) as described below:

* Infliximab;
* Adalimumab;
* Golimumab
* Interferon therapy

Within 8 Weeks of Day 1 [Baseline] (or within 5 half-lives, whichever is longer) and during the study:

* Systemic treatments that could affect vitiligo.
* Use of oral or intravenous immune suppressants (eg, cyclosporine A, tacrolimus, azathioprine, MTX, systemic corticosteroids, mycophenolate-mofetil, mercaptopurine (6MP), or thioguanine).
* Use of sulfasalazine.
* Intralesional, oral or injectable steroids.

Within 6 Weeks of Day 1 (Baseline), during the study, and within 6 weeks of last dose:

- Vaccination with live attenuated, replication-competent vaccine; Current routine household contact with individuals who have been vaccinated with a live attenuated, replication-competent vaccine.

Within 4 weeks (28 Days) of first dose of study intervention or 5 half-lives (if known), whichever is longer and during the study:

* Prohibited CYP3A inducers (see Table 8).
* Herbals that are known to have an effect on drug metabolism.
* Previous administration of investigational drug(s) or vaccines that do not affect vitiligo.

Note: Any investigational or experimental therapy taken, or procedure performed for vitiligo and other autoimmune or immunologic diseases including but not limited to rheumatoid arthritis, psoriasis alopecia areata, thyroid disease, allergic rhinitis, or atopic dermatitis within the previous 1 year should be carefully evaluated. Participants cannot participate in studies of other investigational or experimental therapies or procedures at any time during their participation in this study.

Within 1 Week of Day 1 [Baseline] (or within 5 half-lives, whichever is longer) and during the study:

- Herbal medications with unknown properties or known beneficial effects for vitiligo.

* Prohibited CYP3A substrates as described in Table 8.
* Investigators should consult the SRSD for ritlecitinib for information regarding medication that is prohibited for concomitant use.
* Investigators should consult the product label for any other medication used during the study for information regarding medication that is prohibited for concomitant use.

And 6. Patients suffering from photodermatosis or taking photosensitive drugs, and 7. Patients with more than 33% of leucotrichia on the lesions (Leukotrichia in more than 33% of the face surface area affected with vitiligo lesions OR leukotrichia in more than 33% of the total body surface area affected with vitiligo lesions), and 8. Personal history of skin cancer, and 9. Personal history of any malignancies or a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ will be excluded from the study, and 10. Patients with active infection or other systemic/ inflammatory disease, and 11. Tuberculosis or latent tuberculosis, and 12. Vulnerable people: pregnant or breast-feeding women, minors, adult under guardianship, deprived of freedom or with psychiatric condition, and 13. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation.

14. Participants are excluded from the study if any of the following criteria apply: i. Medical Conditions:

* Any psychiatric condition including recent or active suicidal ideation or behavior that meets any of the following criteria:
* Suicidal ideation associated with actual intent and a method or plan in the past year: "Yes" answers on items 4 or 5 of the C-SSRS administered at the Screening visit (see Appendix 6).
* Previous history of suicidal behaviors in the past 5 years: "Yes" answer (for events that occurred in the past 5 years) to any of the suicidal behavior items of the C-SSRS.
* For adults, any lifetime history of serious suicidal behavior or recurrent suicidal behavior. For adolescents, any previous lifetime history of suicidal behavior.

ii. Medical conditions pertaining to vitiligo and other diseases/conditions affecting the skin:

* Participants that have other types of vitiligo that do not meet criteria for active or stable vitiligo as noted in inclusion criterion #2 (including, but not limited to, segmental vitiligo and mixed vitiligo).
* Currently have active forms of other disorders of pigmentation (including but not limited to Vogt-Koyanagi-Harada disease, malignancy-induced hypopigmentation [melanoma and mycosis fungoides], post-inflammatory hypopigmentation, pityriasis alba [minor manifestation of atopic dermatitis], senile leukoderma [age-related depigmentation], chemical/drug-induced leukoderma, ataxia telangiectasia, tuberous sclerosis, melasma (all types, including mixed), and congenital hypopigmentation disorder including piebaldism, Waardenburg syndrome, hypomelanosis of Ito, incontinentia pigmenti, dyschromatosis symmetrica hereditarian, xeroderma pigmentosum, and nevus depigmentosus). NOTE: Coexistence of halo nevus/nevi (also known as Sutton nevus/nevi) is permitted.
* Currently have active forms of inflammatory skin disease(s) or evidence of skin conditions (for example, morphea, discoid lupus, leprosy, syphilis, psoriasis, seborrheic dermatitis) at the time of the Screening or Baseline Visit that in the opinion of the investigator would interfere with evaluation of vitiligo or response to treatment.
* Have a superficial skin infections within 2 weeks prior to first dose on Day 1. NOTE: participants may be rescreened after the infection resolves.

iii. General Infection History:

* Having a history of systemic infection requiring hospitalization, parenteral antimicrobial, antiviral (including biologic treatment), antiparasitic, antiprotozoal, or antifungal therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1.
* Have active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 1. NOTE: participants may be rescreened after the infection resolves.
* Evidence or history of untreated, currently treated or inadequately treated active or latent infection with Mycobacterium TB as evidenced by the following:
* IGRA test: a positive QFT-G during Screening (completed by central laboratory) or a positive or borderline T-SPOT®TB (performed at local laboratory in Japan, China or those countries where local guidance require T-SPOT®TB testing) during Screening. If the IGRA test results are indeterminate/borderline, the test should be repeated. If the results of the repeat test are indeterminate/borderline, a PPD test may be substituted for the IGRA test only with the approval from the Pfizer medical monitor on a case-by-case basis. (Participants with a history BCG vaccination must have a negative IGRA test).
* A positive QFT-G test or positive or borderline T-SPOT®TB (T-SPOT test) performed within 12 weeks prior to Screening.
* Assessment of the Screening chest imaging for latent or active tuberculosis is required if QFT-G is positive or T-SPOT is positive or borderline or if the participant has been previously treated for latent or active TB and is to be performed according to local standards of care or country-specific guidelines. Chest imaging performed 12 weeks prior to Screening showing no active TB will be accepted with a copy of the report available in the source document.

NOTE: Participants who have previously been adequately treated for latent or active TB (according to WHO/regional or local country recommendations by appropriately qualified personnel as defined by local practice) may be enrolled. Neither a QFT-G test, nor a TSPOT test nor a PPD test is needed provided the treatment, including details of the previous course of therapy (eg, medication(s) used, dose, and duration) is well documented in the participant's medical records and/or source documentation prior to enrollment in the study. A participant who is currently being treated for latent TB infection can only be enrolled with documentation of an adequate treatment regimen that does not include prohibited medications (such as rifamycins [eg, Rifabutin, Rifampin, Rifapentine]), and with prior approval by the sponsor (see Section 8.7).

iv. Specific Viral Infection History:

* History (single episode) of disseminated herpes zoster or disseminated herpes simplex, or a recurrent (more than one episode of) localized, dermatomal herpes zoster.
* Infected with hepatitis B or hepatitis C viruses: all participants will undergo screening for hepatitis B and C for eligibility.
* Hepatitis B: At Screening, hepatitis B surface antigen (HBsAg) and hepatitis B core antibody (HBcAb) will be tested:
* If both tests are negative, the participant is eligible for study inclusion.
* If HBsAg is positive, the participant must be excluded from participation in the study.
* If HBsAg is negative and HBcAb is positive, hepatitis B surface antibody (HBsAb) reflex testing is required:

  1. If HBsAb is negative, the participant must be excluded from participation in the study; OR
  2. If HBsAb is positive, the participant is eligible for study inclusion.
* Hepatitis C: At Screening, hepatitis C antibody (HCVAb) will be tested:
* Participants who are HCVAb negative are eligible.
* Participants who are HCVAb positive will be reflex-tested for hepatitis C (HCV) RNA. Participants who are positive for HCVAb and HCV RNA will not be eligible for this study.
* Have a known immunodeficiency disorder (including positive serology for HIV at Screening) or a first-degree relative with a hereditary immunodeficiency.

  v. Medical Conditions, Other:
* Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (eg, untreated hypovitaminosis D or hypothyroidism), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator or Pfizer (or designee), the participant is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle requirements.

Note: In case hypovitaminosis D (under LLN) is identified for the first time at Screening, treatment should be started at least 7 days prior to baseline.

• History of severe allergic or anaphylactoid reaction to any kinase inhibitor or a known allergy/hypersensitivity to any component (including excipients) of the study intervention.

* Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating or progressive.
* Have a history of any lymphoproliferative disorder such as EBV-related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
* Abnormal findings on the screening chest imaging (eg, chest x-ray) that may increase the risk associated with study participation including, but not limited to, presence of active TB, general infections, cardiomyopathy, or malignancy. Chest imaging may be performed up to 12 weeks prior to Screening. Documentation of the official reading must be located and available in the source documentation.
* Long QT Syndrome, a family history of Long QT Syndrome, or a history of TdP.
* Have any malignancies or have a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
* Significant trauma or major surgery within 1 month of the first dose of study drug or considered in imminent need for surgery or with elective surgery scheduled to occur during the study.

  15. Patients with severe hepatic impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
The Facial Vitiligo Area Scoring Index (F-VASI) | at week 52
  To compare the proportion of patients treated with combined ritlecitinib + nbUVB versus ritlecitinib monotherapy achieving The Facial Vitiligo Area Scoring Index (F-VASI) -75 at week.
Total Body Vitiligo Scoring Index (T-VASI) 50 | at week 52
  To compare the proportion of patients treated with combined ritlecitinib + nbUVB versus ritlecitinib monotherapy achieving T-VASI50 at week 52

SECONDARY OUTCOMES:
Safety treatment | during 52 weeks
  All the adverse events (clinical and biological) occurring over the study period will be collected with their type, grade and severity. At each visit, the investigator will record all the events since the last visit
The quality of life | during 52 weeks
  The quality of life will be assessed by using VIPs (Vitiligo Impact Patient scale) short form at baseline and week 36, week 52 and week 72. VIPs is a transcultural validated specific vitiligo burden tool according to skin phototype. The VIPs-22 which is the latest version of the scale will be used in this study. Evolution will be calculated between baseline and week 36, week 52 and week 72 considering the initial and second randomization to define different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- CHu de Nice, Hôpital Archet, Nice, Alpes-Maritime, France